CLINICAL TRIAL: NCT00923507
Title: Natural History Study of Monoclonal B Cell Lymphocytosis (MBL), Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL), Lymphoplasmacytic Lymphoma (LPL)/Waldenstrom Macroglobulinemia (WM), and Splenic Marginal Zone Lymphoma (SMZL)
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080105; 08-H-0105; NCT00769743 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Monoclonal B-Cell Lymphocytosis; Small Lymphocytic Lymphoma; CLL (Chronic Lymphocytic Leukemia)
Keywords: Chronic Lymphocytic Leukemia (CLL); Monoclonal B Cell Lymphocytosis; Small Lymphocytic Lymphoma (SLL); Natural History; Leukemia; Lymphoma
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with monoclonal B cell lymphocytosis (MBL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), lymphoplasmacytic lymphoma (LPL)/Waldenstr(SqrRoot)(Delta)m macroglobulinemia (WM), and splenic marginal zone lymphoma (SMZL).

SUMMARY:
Background

The development of new technologies now allow scientists to investigate the molecular basis and clinical manifestations of monoclonal B cell lymphocytosis (MBL), chronic lymphocytic leukemia(CLL)/small lymphocytic lymphoma (SLL), lymphoplasmacytic lymphoma (LPL)/Waldenstrom macroglobulinemia (WM), and splenic marginal zone lymphoma (SMZL). Applying these methods in a natural history study can help identify processes involved in disease progression, and possibly lead to the discovery or validation of treatment targets.

Objectives

Study the history of MBL/CLL/SLL/LPL/WM/SMZL in patients prior to and after treatment. Characterize clinical, biologic and molecular events of disease stability and progression of patients enrolled on this protocol.

Eligibility:

* Diagnosis of CLL/SLL and on treatment/previously treated/nearing treatment
* Diagnosis of LPL/WM
* As of February 5, 2025, patients with MBL and SMZL will no longer be enrolled.
* Age greater than or equal to 18 years.
* ECOG performance status of 0-2.

Design

Patients are typically followed every 6 to 24 months in the clinic and have blood drawn. Patients may be asked to undergo additional testing, including bone marrow biopsy and aspiration, lymph node biopsy, positron emission tomography, and CT and MRI scans. Some of these tests (e.g., blood draw) may be required to monitor CLL/SLL and LPL/WM. Other tests (e.g., lymph node biopsy) may not be clinically indicated, but patients may be asked to undergo these procedures for research purposes.

No treatment will be administered on this study. If a patients requires treatment for their cancer, available NIH clinical trials and alternative treatment options will be discussed with the patient.

DETAILED DESCRIPTION:
The purpose of this protocol is to collect blood, tissue (bone marrow and lymph node biopsies) and/or imaging studies (PET and CT scans) from patients with monoclonal B cell lymphocytosis (MBL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), lymphoplasmacytic lymphoma (LPL)/Waldenstrom macroglobulinemia (WM), and splenic marginal zone lymphoma (SMZL).

Assessments will be used for clinical and translational research investigating the molecular basis of MBL, CLL/SLL, LPL/WM, SMZL and their clinical manifestations. New technologies now permit the simultaneous characterization of pathogenic events ranging from the control of gene expression to the characterization of the molecular events of cell-cell interactions. Applying these methods to MBL/CLL/SLL/LPL/WM/SMZL in the context of a natural history protocol can help unravel cellular pathways involved in pathogenesis and disease progression and lead to the discovery or the validation of therapeutic targets. MBL/CLL/SLL/LPL/WM/SMZL is an incurable disease for which there are no reliable cell lines and only a few mouse models. There is an urgent need to obtain a flow of primary samples to advance research into pathogenesis and novel treatment approaches.

Eligibility:

Diagnosis of MBL/CLL/SLL/LPL/WM/SMZL

Age greater than or equal to 18 years.

ECOG performance status of 0-2.

-Design:

Patients will be typically followed every 6-12 months for the first 2 years and every 12-24 months thereafter. Interim visits may occur at the discretion of the research team. Patients may donate cellular products or tissues as appropriate for research purposes. Clinical information will be obtained and stored in a central databank.

* Objectives:

  * Describe the history of MBL/CLL/SLL/WM/SMZL in patients prior to and after treatment.
  * Apply the expertise and available technologies of the investigators to advance our understanding of disease pathogenesis by studying MBL/CLL/SLL and closely related B-cell malignancies, LPL/WM and SMZL
  * Develop novel treatment approaches for CLL/SLL/LPL/WM/SMZL.
  * Provide evaluation, diagnostic studies and monitoring for patients on study.
  * Provide blood and tissue linked to clinical and biologic information for translational studies.
* Endpoints:

  * Treatment-free survival, measured as the time from diagnosis or last therapy to the development of active disease that requires treatment at which time patients will be evaluated for a treatment protocol or seek treatment outside of NIH.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Diagnosis of CLL/SLL will be made according to the updated criteria of the NCI Working Group.

   * on treatment or previously treated
   * requiring or nearing first-line treatment

   OR

   Diagnosis of LPL/WM. LPL is defined as the presence of an intertrabecular pattern of bone marrow infiltration by small lymphocytes showing plasmacytoid/plasma cell differentiation. WM, comprising >95% of LPL cases, describes the clinical syndrome of LPL associated with an IgM monoclonal gammopathy of any concentration. The remaining cases may be IgA, IgM, or non-secreting LPL. Immunophenotyping is required for diagnosis
2. Age greater than or equal to 18 years.
3. ECOG performance status of 0-2.
4. Able to comprehend the investigational nature of the protocol and provide informed consent

EXCLUSION CRITERIA:

1. None

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with monoclonal B cell lymphocytosis (MBL), chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), lymphoplasmacytic lymphoma (LPL)/Waldenstr(SqrRoot)(Delta)m macroglobulinemia (WM), and splenic marginal zone lymphoma (SMZL).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-05-29 (Actual)

PRIMARY OUTCOMES:
Study the natural history of MBL/CLL/SLL in patients prior to the time when their disease requires treatment. | Ongoing
  Treatment free survival, measured as the time from diagnosis or last therapy to the development of active disease that requires treatment at which time patients will be able to change to a treatment protocol or seek treatment outside of NIH.

SECONDARY OUTCOMES:
Characterize clinical, biological and molecular events of disease stability and progression of patients enrolled on this protocol | Ongoing
  Describe the underlying biologic heterogeneity of tumor cells in relation to treatment free survival

CONTACTS AND LOCATIONS:
Overall Officials: Adrian U Wiestner, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Cyr MG, Mhibik M, Qi J, Peng H, Chang J, Gaglione EM, Eik D, Herrick J, Venables T, Novick SJ, Courouble VV, Griffin PR, Wiestner A, Rader C. Patient-derived Siglec-6-targeting antibodies engineered for T-cell recruitment have potential therapeutic utility in chronic lymphocytic leukemia. J Immunother Cancer. 2022 Nov;10(11):e004850. doi: 10.1136/jitc-2022-004850. PMID 36442911
- [Derived] Sun C, Chen YC, Martinez Zurita A, Baptista MJ, Pittaluga S, Liu D, Rosebrock D, Gohil SH, Saba NS, Davies-Hill T, Herman SEM, Getz G, Pirooznia M, Wu CJ, Wiestner A. The immune microenvironment shapes transcriptional and genetic heterogeneity in chronic lymphocytic leukemia. Blood Adv. 2023 Jan 10;7(1):145-158. doi: 10.1182/bloodadvances.2021006941. PMID 35358998
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2008-H-0105.html